CLINICAL TRIAL: NCT02196480
Title: Short and Long-term Immunogenicity and Safety Following the 23-valent Polysaccharide Pneumococcal Vaccine in Juvenile Idiopathic Arthritis Patients Under Anti-TNF Therapy
Brief Title: 23-valent Polysaccharide Pneumococcal Vaccine in Juvenile Idiopathic Arthritis Patients Under Anti-TNF Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Nádia Emi Aikawa, MD, PhD, University of Sao Paulo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PPV23JIA-aTNF
Record Dates: First submitted 2014-07-16; First posted 2014-07-22 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-07

CONDITIONS: Juvenile Idiopathic Arthritis
MeSH Terms: conditions — Arthritis, Juvenile

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Methotrexate (No Intervention): JIA patients on stable dose of methotrexate vaccinated with PPV23
- anti-TNF (Experimental): JIA patients refractory to methotrexate immediately before the association of anti-TNF vaccinated with PPV23
  Interventions: Biological: anti-TNF

INTERVENTIONS:
Biological: anti-TNF — Anti-tumor necrosis factor therapy
  Arms: anti-TNF

SUMMARY:
Objectives: To assess immunogenicity and safety of the 23-valent polysaccharide pneumococcal vaccine (PPV23) in JIA patients with and without anti-TNF therapy. The influences of demographic data, disease activity and treatment on immune response and the potential deleterious effect of vaccine on disease itself were also evaluated.

Methods: 17 JIA patients immediately pre-etanercept (Group 1) and 10 JIA patients on stable dose of methotrexate (Group 2) will receive one dose of PPV23. All patients will be evaluated pre-vaccination, 2 months and 12 months post-vaccination for seven pneumoccocal serotypes. Serology will be performed by enzyme immunoassay and the immunogenicity endpoints will include seroprotection (SP), seroconversion (SP) and geometric mean concentration of antibodies (GMC). Clinical and laboratorial parameters of JIA will be evaluated before and after vaccination.

DETAILED DESCRIPTION:
Seventeen JIA patients (International League Against Rheumatism criteria) followed at the Pediatric Rheumatology Unit of Children's Institute of Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo and who are refractory to methotrexate [median dose 0.9 mg/kg/week (0.7 - 1)] will be included immediately before the association of anti-TNF (etanercept 0.8 mg/kg/week, Group 1) to the previous therapy. The control group (Group 2) consist of 10 JIA patients on stable dose of methotrexate [median dose 0.8 mg/kg/week (0.3-1.0)]. One intramuscular dose of PPV23 (Sanofi Pasteur), lot B0381-3, at the immunization center of the same hospital will be given to each study subject.

Participants are ≥ 5 and ≤ 18 years old and patients with previous vaccination against S. pneumoniae will be excluded. This study was approved by the Local Ethical Committee of our University Hospital and an informed consent was obtained from all participants or their legal guardians.

Vaccine immunogenicity Blood samples will be collected pre-vaccination, 2 months and 12 months post-vaccination for 7 pneumoccocal serotypes (4, 6B, 9V, 14, 18C, 19F, 23F). Samples will be centrifuged and serum will be frozen and stored at -70 ◦C until tested. In order to eliminate non-specific antibodies that may exhibit cross-reactivity, the samples will be pre-absorbed with the C-polysaccharide and with the heterologous serotype 22F.

Serology for each serotype will be performed by enzyme immunoassay and immunogenicity endpoints will include seroprotection rate (SP) (percentage of subjects achieving antibodies titers ≥1.3 micrograms/mL), seroconversion rate (SC) (percentage of subjects with a minimum of 2-fold rise in post-vaccination antibodies titers) and the geometric mean concentration of antibodies (GMC). Adequate vaccine response will be considered when SC occur for at least 50% of all seven vaccine serotypes.

During the period of one year after PPV23 vaccination, all upper and lower respiratory tract infections will be weekly recorded during clinical appointments.

Safety: The number of participants with local and systemic adverse events will be assessed as a measure of safety and tolerability. Local reactions were considered to be related to the PPV23, while systemic adverse events were analyzed individually to determine their causality. Severe adverse events were defined as those requiring hospitalization or death.

Clinical, laboratorial and therapy assessment: All patients will be evaluated on the day of vaccination, 2 months and 12 months after immunization for clinical and laboratorial parameters: number of active joints (swelling within a joint, or limitation in the range of joint movement with joint pain or tenderness), number of limited joints, morning stiffness, patient and physician global assessment of arthritis activity measured with pain scores on the Visual Analog Scale" (VAS) and validated Brazilian version of Childhood Health Assessment Questionnaire (CHAQ). Erythrocyte sedimentation rate (ESR) was evaluated according to Westergreen method and C-reactive protein (CRP) according to nephelometry. The Juvenile Arthritis Disease Activity Score with 27-joint reduced count (JADAS-27), defined as the linear sum of the scores of 4 components [physician global assessment of disease activity (measured on a 10-cm VAS), parent/patient global assessment of well-being (measured on a 10-cm VAS); number of active joints (0-27 joints); and ESR] (range: 0 - 57 points), will be calculated in all JIA patients. Current concomitant treatment with non-steroidal anti-inflammatory drug, prednisone, methotrexate, leflunomide and cyclosporine will be evaluated.

Statistical analysis: Immunogenicity and safety analyses will be descriptive and data will be presented as number (%) or median (range). The GMCs will be compared between JIA patients with and without anti-TNF therapy using a two-sided Student's t-test or Mann-Whitney U-test on the log10-transformed titers. The prospective analysis of GMCs for each of seven pneumococcal serotypes will be performed by Friedman Repeated Measures ANOVA on Ranks. Categorical variables (rates of seroprotection and seroconversion, prednisone and immunosuppressive drugs use) will be compared using Fisher's exact test. The prospective analysis of seroprotection and seroconversion rates for each of seven pneumococcal serotypes will be performed by McNemar's Test. The effects before and after vaccination on disease activity will be analyzed with the Wilcoxon signed ranks test. The statistical significance was set at p value < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Juvenile idiopathic arthritis criteria (International League Against Rheumatism criteria)
* ≥ 5 and ≤ 18 years old

Exclusion Criteria:

* Previous vaccination against S. pneumoniae

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 27 (Actual)
Dates: Start 2008-01; Primary Completion 2011-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Seroprotection rate | 2 months after vacccination
  Sseroprotection rate (SP): percentage of subjects achieving antibodies titers ≥1.3 micrograms/mL
Seroconversion rate | 2 months after vaccination
  Seroconversion rate (SC): percentage of subjects with a minimum of 2-fold rise in post-vaccination antibodies titers
Number of participants with local and systemic adverse events | Until 12 months
  Local reactions were considered to be related to the PPV23, while systemic adverse events were analyzed individually to determine their causality. Severe adverse events were defined as those requiring hospitalization or death.

SECONDARY OUTCOMES:
Seroprotection rate | 12 months after vaccination
  Seroprotection rate (SP): percentage of subjects achieving antibodies titers ≥1.3 micrograms/mL
Seroconversion rate | 12 months after vaccination
  Seroconversion rate (SC): percentage of subjects with a minimum of 2-fold rise in post-vaccination antibodies titers
Juvenile Arthritis Disease Activity Score with 27-joint reduced count (JADAS-27) | 2 months after vaccination
  The Juvenile Arthritis Disease Activity Score with 27-joint reduced count (JADAS-27) is defined as the linear sum of the scores of 4 components [physician global assessment of disease activity (measured on a 10-cm VAS), parent/patient global assessment of well-being (measured on a 10-cm VAS); number of active joints (0-27 joints); and ESR] (range: 0 - 57 points)
Juvenile Arthritis Disease Activity Score with 27-joint reduced count (JADAS-27) | 12 months after vaccination
  The Juvenile Arthritis Disease Activity Score with 27-joint reduced count (JADAS-27) is defined as the linear sum of the scores of 4 components [physician global assessment of disease activity (measured on a 10-cm VAS), parent/patient global assessment of well-being (measured on a 10-cm VAS); number of active joints (0-27 joints); and ESR] (range: 0 - 57 points)

CONTACTS AND LOCATIONS:
Overall Officials: Nadia E Aikawa, MD, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Centro de Dispensação de Medicamentos de Alto Custo (CEDMAC), São Paulo, São Paulo, Brazil